CLINICAL TRIAL: NCT03204032
Title: A Phase II Randomized,Controlled,Open Label,Multicentre Study of Tegafur Combined With Temozolomide Versus Tegafur Combined With Temozolomide and Thalidomide in Subjects With Advanced Extrapancreatic Neuroendocrine Tumor
Brief Title: A Study of Tegafur Combined With Temozolomide Versus Tegafur Combined With Temozolomide and Thalidomide in Subjects With Advanced Extrapancreatic Neuroendocrine Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, Assistant Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-104
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Extrapancreatic Neuroendocrine Tumor
Keywords: Tegafur; Temozolomide; Thalidomide; Extrapancreatic Neuroendocrine Tumor
MeSH Terms: interventions — Tegafur; Temozolomide; Thalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegafur and Temozolomide (Experimental)
  Interventions: Drug: Tegafur; Drug: Temozolomide
- Tegafur and Temozolomide combined with Thalidomide (Active Comparator)
  Interventions: Drug: Tegafur; Drug: Temozolomide; Drug: Thalidomide

INTERVENTIONS:
Drug: Tegafur — Tegafur 40-60mg po bid(d1-d14);
Drug: Temozolomide — 200mg po qd(d10-d14)
Drug: Thalidomide — Thalidomide 100mg po qd(d1-d7) Thalidomide 200mg po qd(d8-d14) Thalidomide 300mg po qd(d15-d21)
  Arms: Tegafur and Temozolomide combined with Thalidomide

SUMMARY:
A Phase II Randomized,Controlled,Open Label,Multicentre Study to evaluate the efficacy and safety of Tegafur combined with Temozolomide versus Tegafur combined with Temozolomide and Thalidomide in subjects with Advanced Extrapancreatic Neuroendocrine Tumor

ELIGIBILITY:
Inclusion Criteria:

1. Patients should participate in the study voluntarily and sign informed consent;
2. Histopathological proven diagnosis of low and intermediate grade (G1, G2 or G3) advanced Extrapancreatic neuroendocrine tumor( locally advanced, unresectable or distant Metastatic). For gastroenteropancreatic neuroendocrine tumor（GEP-NET）,the

   - Page 4 of 5 [DRAFT] - classification is based on nuclear mitotic number and the Ki-67 index,which are as follows:G1:Nuclear mitotic number <2/10HPF,Ki-67 proliferative index ≤2%.G2: Nuclear mitotic number 2～20/10HPF,Ki-67 proliferative index 3%～20%.G3 Nuclear mitotic number > 20/10HPF,Ki-67 proliferative index >20%;
3. Patients with advanced Extrapancreatic neuroendocrine tumor who had not been treated or had no more than two kinds of Systemic Anti-tumor Therapy,which could be somatostatin analogs, interferon, PRRT (peptide receptor radionuclide therapy), mTOR inhibitors, or chemotherapy (without any use of azole amines, fluorouracil,or thalidomide chemotherapy drugs);
4. Radiological documentation of tumor progression is required within 12months prior to randomization;
5. At least one measurable lesion (byRECIST1.1);
6. ANC≥1.5×109/L,PLT≥100×109/L,HB≥90g/L,TBIL≤1.5ULN ;Without supportive care, ALT≤2.5ULN and ALP≤2.5ULN (without hepatic metastasis) ALT≤5ULN and ALP≤5ULN(with hepatic metastasis);serum creatin ≤1.5ULN and creatinine clearance rate

   ≥60ml/min；INR≤1.5ULN and APTT ≤1.5ULN ;
7. ECOG PS:0-1;
8. Life expectancy of more than 12 weeks;
9. Men/Women of childbearing potential must agree to use a highly effective contraceptive method (such as double barrier contraceptive method，condom, oral or injectable contraceptives and intrauterine device) throughout treatment and for at least 90 days after study completion；All female patients will be considered fertile unless she has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexal resection, or radioactive ovarian irradiation etc.)

Exclusion Criteria:

* 1、Diagnosed with high grade (G3) neuroendocrine carcinomas, adenocarcinoma, pancreatic islet cell carcinoma, goblet cell carcinoid, large cell neuroendocrine carcinoma, and small cell carcinoma; 2、Functional NET which needs concomiant use of long-acting somatostatin analogues to control symptoms such as insulinoma, gastrinoma, glucagon tumor, somatostatin, ACTH tumor, VIP tumor, and carcinoid syndrome, Zollinger-Ellison syndrome or other disease-specific active symptoms.

  3、Have received anti-vascular endothelial growth factor（VEGF）/VEGFR targeted drugs and progressed upon these drugs 4、Urinalysis shows urine protein ≥ 2+ or 24-hour protein quantity test shows urinary protein ≥1 g; 5、Serum potassium, calcium (albumin-bound ionic or corrected) or magnesium exceed the normal range with clinical significance； 6、Under anti-hypertension treatment, still uncontrolled hypertension, defined as: systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg; 7、Gastrointestinal disease or condition that investigators suspect may affect drug absorption, including, but not limited to, active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation by investigator's discretion; 8、History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or a thromboembolic event (including transient ischemic attack) within 12 months; 9、Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris or coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; LVEF (LVEF) <50%; 10、Mean corrected QT interval (QTc) ≥ 480 msec; 11、Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection; 12、Anti-tumor therapy received within 4 weeks prior to the initiation of the investigational treatment, including, but not limited to, chemotherapy, radical radiotherapy, targeted therapy, immunotherapy and anti-tumor Chinese medicine treatment, hepatic chemoembolization, cryoablation and radiofrequency ablation ; 13、Palliative radiotherapy for a bone metastasis lesion within 2 weeks prior to the initiation of the investigational treatment; 14、Any clinically significant active infection, including, but not limited to, human immunodeficiency virus (HIV) infection; 15、History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known Hepatitis C virus （HCV) infection with HCV RNA positive (copies ≥1×103/m); or liver cirrhosis, etc.

  16、Surgery (except biopsy) within 28 days prior to the initiation of investigational treatment or unhealed surgical incision; 17、Brain metastases and/or spinal cord compression not treated by surgery and/or radiotherapy, and with no clinical imaging evidence of disease stability; 18、Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for hair loss);

  19、Received investigational treatments in other clinical studies within 4 weeks prior to enrollment; 20、Women who are pregnant or lactating; 21、Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions are inappropriate for the use of the investigational product or affect interpretation of study results.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From randomization，each 6 weeks or 12 weeks(a year later) up to intolerance to the toxicity or PD (up to 24 months)

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | From randomization，each 6 weeks or 12 weeks(a year later) up to intolerable toxicity or PD (up to 24 months)
Time to Tumor Response (TTR) | From randomization，each 6 weeks or 12 weeks(a year later)up to PD or death(up to 24 months)
Duration of Response(DOR) | From randomization，each 6 weeks or 12 weeks(a year later) up to PD or death(up to 24 months)
Progression free survival(PFS) | From randomization，each 6 weeks or 12 weeks(a year later)(a year later) up to PD or death (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chi Y, Song L, Liu W, Zhou Y, Miao Y, Fang W, Tan H, Shi S, Jiang H, Xu J, Jia R, Zheng B, Jiang L, Zhao J, Zhang R, Tan H, Wang Y, Chen Q, Yang M, Guo X, Tong Z, Qi Z, Zhao F, Yan X, Zhao H. S-1/temozolomide versus S-1/temozolomide plus thalidomide in advanced pancreatic and non-pancreatic neuroendocrine tumours (STEM): A randomised, open-label, multicentre phase 2 trial. EClinicalMedicine. 2022 Sep 26;54:101667. doi: 10.1016/j.eclinm.2022.101667. eCollection 2022 Dec. PMID 36188432